CLINICAL TRIAL: NCT00079508
Title: A Phase III Study of Angiomax (Bivalirudin) in Patients With HIT/HITTS Type II Undergoing Cardiac Surgery on Cardiopulmonary Bypass (CPB)
Brief Title: Angiomax in Patients With HIT/HITTS Type II Undergoing CPB
Acronym: HIT/TS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMC-BIV-02-03; CHOOSE-On
Record Dates: First submitted 2004-03-09; First posted 2004-03-11 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Cardiovascular Disease; Coronary Artery Bypass Surgery
Keywords: Heparin-induced Thrombocytopenia; Heparin-induced Thrombocytopenia/Thrombosis Syndrome; HIT/HITTS; Heparin anti-body positive
MeSH Terms: conditions — Cardiovascular Diseases | interventions — bivalirudin

INTERVENTIONS:
Drug: Angiomax (bivalirudin) — 250 mg vial administered as 1.0 mg/kg intravenous (IV) bolus and 2.5 mg/kg/h IV infusion during the procedure with the option to administer additional 0.1 to 0.5 mg/kg boluses to increase the level of anticoagulation as clinically indicated. A low-dose infusion could have been administered in the preoperative phase (up to 48 hours before the procedure) and in the postoperative phase (up to 14 days after the procedure) as clinically indicated for management of HIT/TS. A starting bolus of 0.1 mg/kg and/or an infusion of 0.2 mg/kg/h titrated to a desired activated partial thromboplastin time (aPTT), eg, 1.5-2.5 times baseline aPTT, was recommended.

SUMMARY:
The purpose of this study is to demonstrate that in patients with heparin-induced thrombocytopenia (HIT)/heparin-induced thrombocytopenia and thrombosis syndrome (HITTS) Type II undergoing cardiac surgery on cardiopulmonary bypass (CPB), Angiomax is a safe and effective anticoagulant.

DETAILED DESCRIPTION:
An open-label, prospective, multicenter, single-arm study; with a historical reference cohort of similarly identified HIT/HITTS patients from participating institutions that underwent cardiac surgery on CPB with alternative anticoagulation regimens during the period of approximately 12 months prior to initiation of the first patient into this study.

ELIGIBILITY:
Inclusion Criteria

* Provide written informed consent before initiation of any study-related procedures, and
* Be at least 18 years of age, and
* Be scheduled for CABG, CABG single valve surgery, or isolated single valve surgery on CPB. Patients undergoing repeat (redo) CABG are also considered eligible for this study, and demonstrated
* New diagnosis or history of objectively documented HIT/HITTS Type II, defined as one or more of the following:

  1. Positive heparin-induced platelet aggregation (HIPA) or other functional assay for HIT or immunoassay for HIT antibodies (ELISA), AND/OR
  2. HIT: Thrombocytopenia associated with heparin therapy, where the platelet count has decreased by 50%*, OR
  3. HITTS: Thrombocytopenia (as defined in B above) PLUS any evidence of arterial or venous thrombosis

Exclusion Criteria

* Confirmed pregnancy at time of enrollment via IVRS (if woman of child-bearing potential) (Urine or serum pregnancy test)
* Cerebrovascular accident within 6 months, or any cerebrovascular accident with a residual neurological deficit.
* Intracranial neoplasm, arteriovenous malformation or aneurysm.
* Dependency on renal dialysis or creatinine clearance <30mL/min.
* Ongoing treatment with warfarin (or other oral anticoagulant) at the time of enrollment.

Patients previously treated with warfarin may be enrolled if warfarin therapy can be safely discontinued and baseline INR is < 1.3 times control in the absence of heparin therapy.

* Known allergy to Angiomax or hirudin derived drugs, or known sensitivity to any component of the product.
* Patients receiving clopidogrel (Plavix®) within the previous 5 days may be enrolled if in the opinion of the Investigator the benefits of surgery outweigh the risk associated with recent clopidogrel administration.
* Patients receiving a glycoprotein IIb/IIIa inhibitor within the previous 48 hours prior to enrollment if abciximab (ReoPro®) or 12 hours if eptifibatide (Integrilin®) or tirofiban (Aggrastat®), may be enrolled if in the opinion of the Investigator the benefits of surgery outweigh the risk associated with not waiting the 48 or 12 hour time period prior to enrollment.
* Patients receiving lepirudin (Refludan®) or argatroban within the previous 24 hours prior to enrollment.

Patients currently receiving lepirudin or argatroban can be enrolled if they are switched to Angiomax at least 24 hours prior to the planned cardiac surgery.

* Patients receiving LMWH or thrombolytics within the previous 12 hours may be enrolled if in the opinion of the Investigator the benefits of surgery outweigh the risk associated with not waiting the 12 hour time period.
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment.
* Refusal to undergo blood transfusion should it become necessary.
* Any other disease or condition, which, in the judgment of the Investigator, would place a patient at undue risk by being enrolled in the trial, or cause inability to comply with the trial.
* Planned surgical procedure in which proximal anastomoses will precede distal anastomoses of the bypass grafts.
* Planned (>1) double (or greater) valve repair-replacement (e.g.: AVR-MVR) surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2004-04; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | 7 days
  In-hospital acute procedural success, defined as the absence of death, Q wave MI, repeat coronary revascularization, and stroke (hemorrhagic or ischemic) at hospital discharge or Day 7 after surgery ('Day 7/discharge'), whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Lloyd, MD, Study Director — The Medicines Company
Locations (1):
- The Cleveland Clinic, Cleveland, Ohio, United States